CLINICAL TRIAL: NCT04881942
Title: Characterization of Selected Aerosol Constituents Levels in the Exhaled Breath of Adult e-Vapor Users During Use of Four e-Vapor Products
Brief Title: Characterization of Selected Aerosol Constituents Levels in the Exhaled Breath of Adult e-Vapor Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altria Client Services LLC (Industry)
Collaborators: Cato Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ALCS-RA-17-06-EV
Record Dates: First submitted 2021-04-26; First posted 2021-05-11 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-02

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: This is an open-label, 4-way crossover study designed to estimate the nicotine, glycerin, propylene glycol, menthol, formaldehyde, acetaldehyde, and acrolein levels in exhaled breath samples during use of four MarkTen® XL e-vapor products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ABDC (Experimental): Subjects administered 2 menthol and and 2 non-menthol test e-vapor products:
  Product A (XL25F) on Day 1, Product B (XL40CB) on Day 2, Product D (XL40MB) on Day 3 and Product C (XL35WM) on Day 4
  Interventions: Other: e-Vapor Product A; Other: e-Vapor Product B; Other: e-Vapor Product C; Other: e-Vapor Product D
- BCAD (Experimental): Subjects administered 2 menthol and and 2 non-menthol test e-vapor products:
  Product B (XL40CB) on Day 1, Product C (XL35WM) on Day 2, Product A (XL25F) on Day 3 and Product D (XL40MB) on Day 4
  Interventions: Other: e-Vapor Product A; Other: e-Vapor Product B; Other: e-Vapor Product C; Other: e-Vapor Product D
- CDBA (Experimental): Subjects administered 2 menthol and and 2 non-menthol test e-vapor products:
  Product C (XL35WM) on Day 1 Product D (XL40MB) on Day 2, Product B (XL40CB) on Day 3 and Product A (XL25F) on Day 4
  Interventions: Other: e-Vapor Product A; Other: e-Vapor Product B; Other: e-Vapor Product C; Other: e-Vapor Product D
- DACB (Experimental): Subjects administered 2 menthol and and 2 non-menthol test e-vapor products:
  Product D (XL40MB) on Day 1, Product A (XL25F) on Day 2, Product C (XL35WM) on Day 3 and Product B (XL40CB) on Day 4
  Interventions: Other: e-Vapor Product A; Other: e-Vapor Product B; Other: e-Vapor Product C; Other: e-Vapor Product D

INTERVENTIONS:
Other: e-Vapor Product A — e-Vapor product XL25F
  Other Names: MarkTen® XL Fusion [2.5% nicotine by weight {NBW}] formerly marketed by NuMark LLC
Other: e-Vapor Product B — e-Vapor product XL40CB
  Other Names: MarkTen® XL Bold Classic [4.0% NBW] formerly marketed by NuMark LLC
Other: e-Vapor Product C — e-Vapor product XL35WM
  Other Names: MarkTen® XL Winter Mint [3.5% NBW] formerly marketed by NuMark LLC
Other: e-Vapor Product D — e-Vapor product XL40MB
  Other Names: MarkTen® XL Bold Menthol [4.0% NBW] formerly marketed by NuMark LLC

SUMMARY:
This is an open-label, 4-way crossover study designed to estimate the nicotine, glycerin, propylene glycol, menthol, formaldehyde, acetaldehyde, and acrolein levels in exhaled breath samples during use of four MarkTen® XL e-vapor products. The study will enroll approximately 32 adult e-vapor-using subjects at one site in the United States in High Point, NC.

DETAILED DESCRIPTION:
This is an open-label, 4-way crossover study designed to estimate the nicotine, glycerin, propylene glycol, menthol, formaldehyde, acetaldehyde, and acrolein levels in exhaled breath samples during use of four MarkTen® XL e-vapor products (which are no longer manufactured or sold commercially). The study will enroll approximately 32 adult e-vapor-using (with no more that 60% of either sex). Each of the 32 subjects will provide two exhaled breath samples (10 puffs for each sample) for all four test products. Subjects will make two visits to the site, one screening visit and one 4 day in-clinic visit to provide exhalation samples for four test products (one each day for 4 days). Subjects will also use their assigned test product ad libitum for 12 hours each day after the collection of exhaled breath samples. Subjects will be randomly assigned to a test product-use schedule at Visit 2, with one test product used per day. The anticipated study duration for each subject from screening through completion of all study participation will be approximately 34 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject candidates must satisfy the following criteria before being enrolled in the study:

  1. provide voluntary consent to participate, as documented by the signed institutional review board (IRB)-approved informed consent form (ICF) for the study;
  2. be between the ages of 21 and 65 years, inclusive, at the time of screening (Visit 1);
  3. be positive for tobacco use by urine cotinine measurement (≥ 500 ng/mL) at Visit 1 (screening);
  4. have used nicotine-containing EVPs for the 3 months before Visit 1 (screening) and use of nicotine-containing EVPs ("some days" or "every day") for the past 30 days and at least 4 out of the past 7 days before Visit 1 (screening) and at check-in for Visit 2;
  5. have negative alcohol, amphetamines, opiates, cannabinoids, phencyclidine, and cocaine urine drug screening results (exhaled breath test for alcohol is also acceptable) at Visit 1 (screening) and at check-in for Visit 2;
  6. if female (all females), have a negative serum pregnancy test at Visit 1 (screening) and have a negative urine pregnancy test at check-in for Visit 2;
  7. if female and heterosexually active and of childbearing potential (e.g., not surgically sterile [i.e., bilateral tubal ligation, hysterectomy, or bilateral oophorectomy] at least 6 months before Visit 1 [screening] or at least 2 years naturally postmenopausal [follicle-stimulating hormone ≥40 IU/L at Visit 1 (screening)]), must be using one of the following forms of contraception and agree to continue using it through at least 30 days after the last study product use (if early terminated) or completion of the study:

     * hormonal (e.g., oral, transdermal patch, implant, or injection) consistently for at least 3 months before Visit 1 (screening);
     * double barrier (i.e., condom with spermicide or diaphragm with spermicide) consistently for at least 30 days before Visit 1 (screening);
     * intrauterine device for at least 3 months before Visit 1 (screening);
     * Essure® or similar nonsurgical sterilization procedure at least 3 months before Visit 1 (screening); or
     * partner who has been vasectomized for at least 6 months (inclusive) before Visit 1 (screening);
  8. if male and heterosexually active and capable of fathering a child (e.g., not vasectomized at least 6 months before Visit 1 [screening]), must be using a double barrier (i.e., condom with spermicide or diaphragm with spermicide) method of contraception from check-in at Visit 2 until at least 90 days after the last study product use (if early terminated) or completion of the study;
  9. not plan to quit e-vapor use in the next 30 days;
  10. be willing to use all assigned EVPs during the study; and
  11. be willing and able to comply with the requirements of the study.

Exclusion Criteria:

* Subjects may be excluded from the study if the subject meets any of the criteria listed below at Visit 1 (screening) and Visit 2 or at any time during the study as appropriate. Exceptions may be permitted at the discretion of the investigator in consultation with the Sponsor, providing there would be no additional risk involved for the subject. Any exceptions will be documented.

  1. have a history or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, diabetes, existing respiratory diseases (especially bronchospastic diseases and asthma), immunologic, psychiatric, cardiovascular disease, or any other condition(s) that, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results (Note: Chronic medical conditions controlled and on stable medications [over the past 3 months] may not be exclusionary per investigator discretion);
  2. have current evidence or any history of congestive heart failure;
  3. have clinically significant abnormal findings on physical examination, vital signs, ECG, clinical laboratory results, or medical history, in the opinion of the investigator;
  4. have systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg at Visit 1 (screening) or at check-in for Visit 2;
  5. have estimated creatinine clearance (by Cockcroft-Gault equation) <80 mL/minute;
  6. have liver enzymes (aspartate aminotransferase and alanine aminotransferase) ≥1.5 times the upper limit of normal at Visit 1 (screening);
  7. have an acute illness (e.g., upper respiratory infection or viral infection) requiring treatment within 2 weeks before check-in at Visit 2;
  8. have fever (>100.5°F) at Visit 1 (screening) or at check-in for Visit 2;
  9. have body mass index (BMI) greater than 40.0 kg/m2 or less than 18.0 kg/m2 at Visit 1 (screening);
  10. have positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at Visit 1 (screening);
  11. have used prescription or over-the-counter bronchodilator medication (e.g., inhaled or oral β-agonists) within 12 months of Visit 1 (screening) and Visit 2;
  12. have diabetes mellitus that is not controlled by diet/exercise alone, in the opinion of the investigator;
  13. have used prescription antidiabetic medication or insulin therapy within 12 months of Visit 1 (screening) and Visit 2;
  14. have used medication for depression or asthma within 12 months of Visit 1 (screening) and Visit 2;
  15. have a history of drug or alcohol abuse within 12 months of Visit 1 (screening) and Visit 2;
  16. have had allergic or other known adverse reactions to menthol, propylene glycol, or glycerol;
  17. if female, be pregnant, nursing, or planning to become pregnant during the study;
  18. have participated in a clinical study for an investigational drug, medical device, biologic, or for a tobacco product within 30 days before Visit 1 (screening) and Visit 2;
  19. be a current or former employee of the tobacco industry or a first-degree relative (e.g., parent, spouse, sibling, child) of a current or former employee of the tobacco industry or a named party or class representative in litigation with any tobacco company;
  20. have been involved in the development of the study design/conduct or be a first-degree relative (e.g., parent, spouse, sibling, child) of someone involved in the development of the study design/conduct;
  21. be a current employee or personnel involved with the study at the site; or
  22. have participated in two or more ALCS studies within the past 12-month period before Visit 1 (screening) and check in at Visit 2.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2018-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery S Edmiston, PhD, Study Director — Altria Client Services
Locations (1):
- High Point Clinical Trials Center, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Poster presentation at 2018 Society for Research in Nicotine and Tobacco annual meeting entitled: Exhaled Breath Levels of Selected Constituents From Controlled Use of MarkTen® e-Vapor Products in Adult e-Vapor Users — https://sciences.altria.com/-/media/Project/Altria/Sciences/presentations/2/2018-SRNT--Edmiston-Feb-24-Exhaled-Breath-Levels-of-Selected-Constituents.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 subjects (including alternates) used at least one test product during the Day -1 Trial. One subject discontinued from the study before randomization; 2 alternates were discontinued prior to randomization once the enrollment goal of 32 subjects was met. Therefore, a total of 32 subjects were randomized into the study. The 3 subjects who were discontinued prior to randomization constitute the "Day -1 Trial" group and are included in the Safety Population for AE reporting, and Baseline data.
Groups:
- ABDC: Subjects administered 2 menthol and 2 non-menthol test e-vapor products:
  Product A (XL25F) on Day 1, Product B (XL40CB) on Day 2, Product D (XL40MB) on Day 3 and Product C (XL35WM) on Day 4
- BCAD: Subjects administered 2 menthol and 2 non-menthol test e-vapor products:
  Product B (XL40CB) on Day 1, Product C (XL35WM) on Day 2, Product A (XL25F) on Day 3 and Product D (XL40MB) on Day 4
- CDBA: Subjects administered 2 menthol and 2 non-menthol test e-vapor products:
  Product C (XL35WM) on Day 1 Product D (XL40MB) on Day 2, Product B (XL40CB) on Day 3 and Product A (XL25F) on Day 4
- DACB: Subjects administered 2 menthol and 2 non-menthol test e-vapor products:
  Product D (XL40MB) on Day 1, Product A (XL25F) on Day 2, Product C (XL35WM) on Day 3 and Product B (XL40CB) on Day 4
- Day -1 Trial: Subjects who used at least one test product during the Visit 2, Day -1 product trial, but were not subsequently randomized.
Period: Overall Study
Arm/Group | ABDC | BCAD | CDBA | DACB | Day -1 Trial
Started | 8 | 8 | 8 | 8 | 3
Completed Day 1 Product Use | 8 | 8 | 8 | 8 | 0
Completed Day 2 Product Use | 8 | 8 | 8 | 8 | 0
Completed Day 3 Product Use | 8 | 8 | 8 | 8 | 0
Completed Day 4 Product Use | 8 | 8 | 8 | 8 | 0
Completed | 8 | 8 | 8 | 8 | 0
Not Completed | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Alternates | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Day-1 Trial: Subjects who used at least one test product during the Visit 2, Day -1 product trial, but were not subsequently randomized
- Total: Total of all reporting groups
Arm/Group | ABDC | BCAD | CDBA | DACB | Day-1 Trial | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 3 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 3 | 35
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.3 (12.02) | 34.9 (12.49) | 41.1 (15.95) | 35.4 (11.73) | 37.7 (14.22) | 36.7 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 3 | 1 | 15
  Male | 4 | 4 | 5 | 5 | 2 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 7 | 8 | 8 | 3 | 31
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 5 | 4 | 2 | 24
  White | 1 | 1 | 3 | 4 | 1 | 10
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Annual Household Income [Count of Participants; unit: Participants] — Subject responses to Demographics survey question "What was your annual household income from all sources over the past year?"
  Participants
    <$20,000 | 4 | 3 | 3 | 7 | 1 | 18
    $20,000-$29,999 | 0 | 4 | 2 | 1 | 1 | 8
    $30,000-$39,999 | 1 | 1 | 1 | 0 | 0 | 3
    $40,000-$49,999 | 1 | 0 | 1 | 0 | 0 | 2
    $50,000-$59,999 | 0 | 0 | 1 | 0 | 0 | 1
    $75,000-$99,999 | 1 | 0 | 0 | 0 | 0 | 1
    No answer | 1 | 0 | 0 | 0 | 1 | 2
Education [Count of Participants; unit: Participants] — Subject responses to Demographics survey question "What is the highest grade or year of school you completed?"
  Participants
    9-11 years | 0 | 0 | 0 | 1 | 1 | 2
    12 years or GED | 2 | 3 | 3 | 4 | 1 | 13
    Some college | 3 | 4 | 3 | 3 | 1 | 14
    College graduate | 1 | 1 | 2 | 0 | 0 | 4
    Other | 1 | 0 | 0 | 0 | 0 | 1
    No answer | 1 | 0 | 0 | 0 | 0 | 1
Height [Mean (Standard Deviation); unit: cm] — Summary of subject height (in cm) by Sequence
  cm | 168.6 (8.16) | 174.6 (7.99) | 170.7 (10.28) | 172.7 (8.40) | 177.7 (22.64) | 172.1 (10.04)
Weight [Mean (Standard Deviation); unit: kg] — Summary of subject weight (in kg) by Sequence
  kg | 80.4 (17.90) | 91.3 (21.44) | 82.8 (11.91) | 76.0 (19.60) | 77.1 (11.46) | 82.1 (17.56)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] — Summary of Subject BMI (in kg/m2) by Sequence
  kg/m² | 28.16 (5.535) | 29.89 (6.014) | 28.48 (3.699) | 25.26 (5.177) | 24.97 (6.035) | 27.69 (5.254)
Employment Status [Count of Participants; unit: Participants]
  Wage Earner | 2 | 6 | 3 | 3 | 2 | 16
  Self-Employed | 1 | 1 | 2 | 1 | 0 | 5
  Unemployed > 1 year | 1 | 0 | 1 | 0 | 0 | 2
  Unemployed < 1 year | 2 | 0 | 1 | 0 | 0 | 3
  Homemaker | 2 | 0 | 0 | 1 | 0 | 3
  Student | 0 | 1 | 0 | 2 | 0 | 3
  Retired | 0 | 0 | 1 | 0 | 0 | 1
  Unable to work | 0 | 0 | 0 | 1 | 1 | 2
Military Experience [Count of Participants; unit: Participants]
  Active Duty | 1 | 0 | 0 | 0 | 0 | 1
  Discharged More Than 1 Year Ago | 1 | 0 | 0 | 1 | 0 | 2
  Never in military | 6 | 7 | 8 | 7 | 3 | 31
  No answer | 0 | 1 | 0 | 0 | 0 | 1
Marital Status [Count of Participants; unit: Participants]
  Single | 5 | 4 | 6 | 6 | 2 | 23
  Married/Partnered | 1 | 2 | 1 | 1 | 0 | 5
  Divorced/Separated/Widowed | 0 | 1 | 1 | 1 | 1 | 4
  No answer | 2 | 1 | 0 | 0 | 0 | 3
Sexual Identity [Count of Participants; unit: Participants]
  Heterosexual or Straight | 7 | 7 | 8 | 8 | 3 | 33
  No answer | 1 | 1 | 0 | 0 | 0 | 2
Previous Cigarette Usage [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "Ever smoked Cigarettes?"
  Participants
    Yes | 7 | 8 | 8 | 8 | 3 | 34
    No | 1 | 0 | 0 | 0 | 0 | 1
100 or more lifetime cigarettes [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "Smoked >= 100 cigarettes in lifetime"
  Participants
    Yes | 6 | 7 | 8 | 8 | 3 | 32
    No | 0 | 1 | 0 | 0 | 0 | 1
    Missing Response / Skip Logics | 2 | 0 | 0 | 0 | 0 | 2
Smoke on a regular basis [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "Ever smoked on regular basis"
  Participants
    Yes | 7 | 7 | 8 | 8 | 3 | 33
    No | 0 | 0 | 0 | 0 | 0 | 0
    Missing Response / Skip Logics | 1 | 1 | 0 | 0 | 0 | 2
Length of Consistent Smoking [Mean (Standard Deviation); unit: Years] — Subject responses were collected from the product-use survey question "How long did you smoke consistently?" Population: Not all participants were asked to respond due to skip logics.
  Years
    number analyzed (Participants) | 7 | 7 | 8 | 8 | 3 | 33
    (all) | 9.9 (8.23) | 12.7 (9.69) | 19.1 (14.70) | 13.0 (13.90) | 13.7 (7.09) | 13.8 (11.57)
Smoking Frequency in past 30 days [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "How often did you smoke in the past 30 days?"
  Participants
    Every Day | 4 | 4 | 3 | 1 | 1 | 13
    Some Days | 2 | 1 | 2 | 3 | 1 | 9
    Not at all | 1 | 2 | 3 | 4 | 1 | 11
    Missing Response / Skip Logics | 1 | 1 | 0 | 0 | 0 | 2
Daily Cigarette Use [Mean (Standard Deviation); unit: number of cigarettes] — Subject responses were collected from the product-use survey question "In the past 30 days how many cigarettes did you smoke per day?". Population: Based on each subject's smoking history, not all subjects were required to answer this question.
  number of cigarettes
    number analyzed (Participants) | 6 | 5 | 5 | 4 | 2 | 22
    (all) | 9.7 (5.96) | 9.0 (4.30) | 9.6 (5.55) | 2.8 (2.22) | 14.0 (8.49) | 8.6 (5.64)
Menthol Cigarettes Regularly [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "Are the cigarettes that you regularly smoke, menthol?"
  Participants
    Yes | 6 | 4 | 4 | 3 | 2 | 19
    No | 0 | 1 | 1 | 1 | 0 | 3
    Missing Response / Skip Logics | 2 | 3 | 3 | 4 | 1 | 13
Daily Smoking [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "Have you smoked daily (or nearly so) during the last year?"
  Participants
    Yes | 4 | 4 | 5 | 2 | 1 | 16
    No | 2 | 1 | 0 | 2 | 1 | 6
    Missing Response / Skip Logics | 2 | 3 | 3 | 4 | 1 | 13
Previously Quit Smoking [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "Have you quit smoking for at least 1 day during the last year?"
  Participants
    Yes | 2 | 2 | 1 | 1 | 1 | 7
    No | 4 | 3 | 4 | 3 | 1 | 15
    Missing Response / Skip Logics | 2 | 3 | 3 | 4 | 1 | 13
Quit Smoking Completely [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "Have you quit smoking completely?"
  Participants
    Yes | 1 | 2 | 3 | 4 | 0 | 10
    No | 6 | 5 | 5 | 4 | 3 | 23
    Missing Response / Skip Logics | 1 | 1 | 0 | 0 | 0 | 2
Current Quit Smoking Duration [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "How long have you quit smoking (currently)?"
  Participants
    < 6 months | 0 | 0 | 0 | 1 | 0 | 1
    > 6 months | 1 | 2 | 3 | 3 | 0 | 9
    Missing Response / Skip Logics | 7 | 6 | 5 | 4 | 3 | 25
Previous E-Cigarette Usage [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "Have you ever tried an e-cigarette?"
  Participants
    Yes | 8 | 8 | 8 | 8 | 3 | 35
    No | 0 | 0 | 0 | 0 | 0 | 0
Type of e-Cigarette and e-Vapor Product Use [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "What types of e-cigarette and e-vapor products do you currently use?". Type 1 = Disposable e-cigarettes; Type 2 = Rechargeable e-cigarettes with pre-filled cartridges that are replaced; Type 3 = Any type of rechargeable e-cigarette or e-vapor product that you refill with e-liquid
  Participants
    Type 1 | 2 | 0 | 0 | 1 | 1 | 4
    Type 2 | 1 | 4 | 2 | 0 | 1 | 8
    Type 3 | 4 | 2 | 5 | 6 | 0 | 17
    Type 1 + Type 2 | 0 | 0 | 1 | 0 | 0 | 1
    Type 1 + Type 3 | 1 | 1 | 0 | 0 | 0 | 2
    Type 2 + Type 3 | 0 | 0 | 0 | 1 | 1 | 2
    Type 1 + Type 2 + Type 3 | 0 | 1 | 0 | 0 | 0 | 1
Number of Days of e-cigarette Use in Past Week [Mean (Standard Deviation); unit: days] — Subject responses were collected from the product-use survey question "In the last week how many days did you use an e-cigarette?"
  days | 6.0 (1.20) | 6.6 (0.74) | 6.6 (1.06) | 6.8 (0.46) | 7.0 (0.00) | 6.5 (0.89)
30 Day Disposable E-Cigarette/Cartridge Count [Mean (Standard Deviation); unit: E-Cigarettes/Cartridges] — Subject responses were collected from the product-use survey question "In the last 30 days how many disposable e-cigarettes or cartridges did you use?"
  E-Cigarettes/Cartridges | 0.6 (0.74) | 0.6 (0.74) | 0.3 (0.46) | 0.9 (1.64) | 3.7 (5.51) | 0.9 (1.85)
Milliliters of E-Liquid/day in last 30 Days [Mean (Standard Deviation); unit: ml/day] — Subject responses were collected from the product-use survey question "In the last 30 days how many mls e-liquid did you use per day?"
  ml/day | 3.6 (6.72) | 2.1 (3.31) | 4.6 (6.70) | 3.5 (3.12) | 2.0 (3.46) | 3.3 (4.94)
e-Cigarette Length of Use [Mean (Standard Deviation); unit: months] — Subject responses were collected from the product-use survey question "How many months have you been using e-cigarettes?"
  months | 17.8 (10.98) | 14.5 (6.02) | 22.5 (15.96) | 17.8 (8.70) | 11.3 (11.02) | 17.5 (10.90)
e-Cigarette Use Frequency in Past 30 Days [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "How often did you use e-cigarettes in the past 30 days?"
  Participants
    Every Day | 4 | 8 | 6 | 7 | 3 | 28
    Some Days | 4 | 0 | 2 | 1 | 0 | 7
    Not at all | 0 | 0 | 0 | 0 | 0 | 0
Quit E-Cigarettes in Last Year [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "Have you quit using e-cigarettes in the last 12 months?"
  Participants
    Yes | 1 | 0 | 0 | 0 | 0 | 1
    No | 7 | 8 | 8 | 8 | 3 | 34
Plan to Quit Smoking [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "Do you plan to quit smoking in the next 30 days?"
  Participants
    Yes | 1 | 0 | 1 | 2 | 0 | 4
    No | 5 | 5 | 5 | 2 | 3 | 20
    Missing Response / Skip Logics | 2 | 3 | 2 | 4 | 0 | 11
Plan to Quit E-Cigarettes [Count of Participants; unit: Participants] — Subject responses were collected from the product-use survey question "Are you planning to quit using e-cigarettes in the next 30 days?"
  Participants
    Yes | 0 | 0 | 0 | 0 | 0 | 0
    No | 8 | 8 | 8 | 8 | 3 | 35

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Residue Summary Statistics by Test-Product Group
Description: Table summarizes the amount of analyte present in exhaled breath after test product use.
  Analyte was collected over an approximately 10-min collection period in the exhaled breath product use session on day the subject was assigned the indicated test product according to the randomization scheme. In the exhaled breath test product use session, one exhaled breath sample was collected using an empty cartridge and inactive battery [sham condition] followed by an exhaled breath sample using the test product. Each exhaled breath sample was collected separately into the same type of trapping container (capturing the specific analyte). Each sample consisted of all the exhaled breath occurring during 10 puffs, each with 5 second puff duration (+/- 1 sec), over ~5 min (one puff approximately every 30 secs) collected in the respective sample collection containers. Sham-corrected analyte amounts were computed by subtracting corresponding sham response values from test product response values.
Time Frame: Data collected over an approximately 10-minute timeframe (2 consecutive exhaled breath samples of 5-minute durations each) on the day the subject was assigned to use the test product (Day 1 or Day 2 or Day 3 or Day 4 according to the randomization scheme)
Measure: Mean (Standard Deviation); unit: Micrograms
Groups:
- e-Vapor Product A: Product XL25F = Test e-vapor product (EVP) (formerly marketed by Nu Mark LLC as MarkTen® XL Fusion [2.5% nicotine by weight {NBW}])
  e-Vapor Product A: e-Vapor product
- e-Vapor Product B: Product XL40CB = Test EVP (formerly marketed by Nu Mark LLC as MarkTen® XL Bold Classic [4.0% NBW]) e-Vapor Product B: e-Vapor product
- e-Vapor Product C: Product XL35WM = Test EVP (formerly marketed by Nu Mark LLC as MarkTen® XL Winter Mint [3.5% NBW]) e-Vapor Product C: e-Vapor product
- e-Vapor Product D: Product XL40MB = Test EVP (formerly marketed by Nu Mark LLC as MarkTen® XL Bold Menthol [4.0% NBW])
  e-Vapor Product D: e-Vapor product
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 31
Micrograms | 87.1 (120.11) | 192.3 (268.53) | 174.1 (208.64) | 182.8 (253.88)

2. Primary Outcome: Sham Nicotine Residue Summary Statistics by Test-Product Group
Description: Table summarizes the amount of analyte present in exhaled breath after sham.
  The analyte was collected over an approximately 10-min collection period in the exhaled breath product use session on the day the subject was assigned the indicated test product according to the randomization scheme. In the exhaled breath test product use session, one exhaled breath sample was collected using an empty cartridge and inactive battery [sham condition] followed by an exhaled breath sample using the test product. Each exhaled breath sample was collected separately into the same type of trapping container (capturing the specific analyte). Each sample consisted of all the exhaled breath occurring during 10 puffs, each with 5 second puff duration (+/- 1 sec), over ~5 min (one puff approximately every 30 sec) collected in the respective sample collection containers. Sham-corrected analyte amounts were computed by subtracting corresponding sham response values from test product response values.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 0.9 (0.66) | 0.9 (0.66) | 0.9 (0.70) | 0.9 (0.69)

3. Primary Outcome: Total Sham-Corrected Nicotine Summary Statistics by Test Product Group
Description: Table presents difference in total analyte amount in exhaled breath samples between sham (inactive battery & empty cartridge) and controlled test product use.
  Analyte was collected over an approximately 10-min collection period in the exhaled breath product use session on day the subject was assigned the indicated test product. In the exhaled breath test product use session, 1 exhaled breath sample was collected using an empty cartridge & inactive battery [sham condition] followed by an exhaled breath sample using the test product. Each exhaled breath sample was collected separately into the same type of trapping container. Each sample consisted of all the exhaled breath occurring during 10 puffs, each with 5 second puff duration (+/- 1 sec), over ~5 min (one puff approximately every 30 secs) collected in the respective sample collection containers. Sham-corrected analyte amounts were computed by subtracting corresponding sham response values from test product response values.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 31
Micrograms | 86.1 (120.40) | 191.4 (268.78) | 173.1 (208.93) | 181.8 (254.23)
Statistical Analysis 1: Comparison: e-Vapor Product A; Null Hypothesis: Mean sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham) analyte amount is equal to 0. Alternate Hypothesis: Mean sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham) analyte amount is not equal to 0; Test type: Equivalence — Null Hypothesis: Mean sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham) analyte amount is equal to 0. Alternate Hypothesis: Mean sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham) analyte amount is not equal to 0; p = 0.0184, ANCOVA; Mean Difference (Net) = 89.44, 95% CI 2-sided [15.77 to 163.11] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 2: Comparison: e-Vapor Product B; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 195.70, 95% CI 2-sided [122.01 to 269.38] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 3: Comparison: e-Vapor Product C; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 168.83, 95% CI 2-sided [95.17 to 242.50] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 4: Comparison: e-Vapor Product D; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 182.65, 95% CI 2-sided [108.63 to 256.67] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)

4. Primary Outcome: Glycerin Residue Summary Statistics by Test-Product Group
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 31
Micrograms | 5964.4 (5029.33) | 5707.3 (5015.41) | 6516.6 (5387.80) | 5682.4 (5156.04)

5. Primary Outcome: Sham Glycerin Residue Summary Statistics by Test-Product Group
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 15.4 (16.49) | 11.1 (5.01) | 15.4 (16.53) | 10.9 (2.65)

6. Primary Outcome: Total Sham-Corrected Glycerin Summary Statistics by Test Product Group
Description: as for outcome 3
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 31
Micrograms | 5949.0 (5033.63) | 5696.2 (5015.99) | 6501.2 (5385.54) | 5671.5 (5155.84)
Statistical Analysis 1: Comparison: e-Vapor Product A; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 5972.3, 95% CI 2-sided [4191.1 to 7753.6] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 2: Comparison: e-Vapor Product B; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 6099.5, 95% CI 2-sided [4317.8 to 7881.2] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 3: Comparison: e-Vapor Product C; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 6484.7, 95% CI 2-sided [4701.7 to 8267.6] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 4: Comparison: e-Vapor Product D; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 5366.8, 95% CI 2-sided [3575.9 to 7157.7] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)

7. Primary Outcome: Menthol Residue Summary Statistics by Test-Product Group
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 31
Micrograms | 0.4 (0.13) | 0.4 (0.08) | 22.1 (9.99) | 31.3 (15.12)

8. Primary Outcome: Sham Menthol Residue Summary Statistics by Test-Product Group
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 0.5 (0.42) | 0.4 (0.08) | 0.4 (0.08) | 0.4 (0.08)

9. Primary Outcome: Total Sham-Corrected Menthol Summary Statistics by Test Product Group
Description: as for outcome 3
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 31
Micrograms | -0.1 (0.30) | 0.0 (0.00) | 21.7 (9.98) | 30.9 (15.12)
Statistical Analysis 1: Comparison: e-Vapor Product A; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.9150, ANCOVA; Mean Difference (Net) = 0.17, 95% CI 2-sided [-2.92 to 3.25] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham) analyte amount is not equal to 0
Statistical Analysis 2: Comparison: e-Vapor Product B; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.8217, ANCOVA; Mean Difference (Net) = 0.35, 95% CI 2-sided [-2.70 to 3.40] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 3: Comparison: e-Vapor Product C; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 21.11, 95% CI 2-sided [18.06 to 24.16] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: e-Vapor Product D; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 31.01, 95% CI 2-sided [27.91 to 34.12] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)

10. Primary Outcome: Propylene Glycol Residue Summary Statistics by Test-Product Group
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 31
Micrograms | 1697.6 (2351.62) | 1047.7 (1497.14) | 3343.4 (4090.27) | 2675.8 (3794.98)

11. Primary Outcome: Sham Propylene Glycol Residue Summary Statistics by Test-Product Group
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 14.9 (1.54) | 14.9 (2.18) | 15.4 (2.97) | 14.6 (0.66)

12. Primary Outcome: Total Sham-Corrected Propylene Glycol Summary Statistics by Test Product Group
Description: as for outcome 3
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 31
Micrograms | 1682.7 (2351.82) | 1032.8 (1497.42) | 3328.0 (4090.90) | 2661.2 (3795.07)
Statistical Analysis 1: Comparison: e-Vapor Product A; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .0031, ANCOVA; Mean Difference (Net) = 1678.4, 95% CI 2-sided [592.14 to 2764.6] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 2: Comparison: e-Vapor Product B; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .0310, ANCOVA; Mean Difference (Net) = 1199.7, 95% CI 2-sided [113.74 to 2285.7] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 3: Comparison: e-Vapor Product C; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 3354.5, 95% CI 2-sided [2266.6 to 4442.3] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 4: Comparison: e-Vapor Product D; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 2511.0, 95% CI 2-sided [1416.1 to 3605.9] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)

13. Primary Outcome: Formaldehyde Residue Summary Statistics by Test-Product Group
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 1.0 (0.74) | 1.1 (0.95) | 1.3 (0.92) | 1.2 (0.85)

14. Primary Outcome: Sham Formaldehyde Residue Summary Statistics by Test-Product Group
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 0.8 (0.66) | 0.8 (0.63) | 1.0 (0.79) | 1.0 (0.79)

15. Primary Outcome: Total Sham-Corrected Formaldehyde Summary Statistics by Test Product Group
Description: as for outcome 3
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 0.19 (0.241) | 0.33 (0.650) | 0.35 (0.326) | 0.27 (0.329)
Statistical Analysis 1: Comparison: e-Vapor Product A; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = .0002, ANCOVA; Mean Difference (Net) = 0.25, 95% CI 2-sided [0.12 to 0.38] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: e-Vapor Product B; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.0003, ANCOVA; Mean Difference (Net) = 0.25, 95% CI 2-sided [0.12 to 0.38] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 3: Comparison: e-Vapor Product C; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 0.34, 95% CI 2-sided [0.21 to 0.47] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)
Statistical Analysis 4: Comparison: e-Vapor Product D; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 0.30, 95% CI 2-sided [0.17 to 0.43] — Mean value is sham-corrected (amount of analyte in test-product exhale minus analyte concentration in exhaled sham)

16. Primary Outcome: Acetaldehyde Residue Summary Statistics by Test-Product Group
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 0.50 (0.000) | 0.50 (0.000) | 0.50 (0.000) | 0.50 (0.000)

17. Primary Outcome: Sham Acetaldehyde Residue Summary Statistics by Test-Product Group
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 0.50 (0.000) | 0.50 (0.000) | 0.50 (0.000) | 0.50 (0.000)

18. Primary Outcome: Total Sham-Corrected Acetaldehyde Summary Statistics by Test Product Group
Description: as for outcome 3
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

19. Primary Outcome: Acrolein Residue Summary Statistics by Test-Product Group
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 0.63 (0.000) | 0.63 (0.000) | 0.63 (0.000) | 0.63 (0.000)

20. Primary Outcome: Sham Acrolein Residue Summary Statistics by Test-Product Group
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 0.6 (0.00) | 0.6 (0.00) | 0.6 (0.00) | 0.6 (0.00)

21. Primary Outcome: Total Sham-Corrected Acrolein Summary Statistics by Test Product Group
Description: as for outcome 3
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: Micrograms
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Micrograms | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

22. Secondary Outcome: Cartridge Weight (g) Change Summary Statistics for Sample 1 (Propylene Glycol, Glycerin, Nicotine, Menthol) by Test Product in the Exhaled-Breath Sessions
Description: Difference in recorded weight of Sample 1, measured in grams, collected before and after product use in Exhaled Breath Sessions. Sample 1 was used to collect propylene glycol, glycerin, nicotine and menthol, and was collected approximately 1 hour before Sample 2.
Time Frame: Samples collected during the approximately 1 hour controlled exhaled breath product use session on the day the subject was assigned to use the test product (Day 1 or Day 2 or Day 3 or Day 4 according to the randomization scheme)
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Grams | 0.0352 (0.008701) | 0.0337 (0.011374) | 0.0402 (0.012596) | 0.0367 (0.012324)
Statistical Analysis 1: Comparison: e-Vapor Product A; Null Hypothesis: Mean cartridge weight change is equal to 0. Alternate Hypothesis: Mean cartridge weight change is not equal to 0; Test type: Equivalence — Null Hypothesis: Mean cartridge weight change is equal to 0. Alternate Hypothesis: Mean cartridge weight change is not equal to 0; p < .0001, ANOVA; Mean Difference (Final Values) = 0.035, 95% CI 2-sided [0.031 to 0.039]
Statistical Analysis 2: Comparison: e-Vapor Product B; [analysis description as in outcome 22, analysis 1]; Test type: Equivalence — [test comment as in outcome 22, analysis 1]; p < .0001, ANOVA; Mean Difference (Net) = 0.034, 95% CI 2-sided [0.030 to 0.038]
Statistical Analysis 3: Comparison: e-Vapor Product C; [analysis description as in outcome 22, analysis 1]; Test type: Equivalence — [test comment as in outcome 22, analysis 1]; p < .0001, ANOVA; Mean Difference (Net) = 0.040, 95% CI 2-sided [0.036 to 0.044]
Statistical Analysis 4: Comparison: e-Vapor Product D; [analysis description as in outcome 22, analysis 1]; Test type: Equivalence — [test comment as in outcome 22, analysis 1]; p < .0001, ANOVA; Mean Difference (Net) = 0.037, 95% CI 2-sided [0.033 to 0.041]

23. Secondary Outcome: Cartridge Weight (g) Change Summary Statistics for Sample 2 (Formaldehyde, Acetaldehyde, Acrolein) by Test Product in the Exhaled-Breath Sessions
Description: Difference in recorded weight of Sample 2, measured in grams, collected before and after product use in Exhaled Breath Sessions, Sample 2 was used to collect formaldehyde, acetaldehyde and acrolein, and was collected approximately 1 hour after Sample 1.
Time Frame: as for outcome 22
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Grams | 0.0356 (0.011530) | 0.0363 (0.011936) | 0.0412 (0.014581) | 0.0379 (0.012395)
Statistical Analysis 1: Comparison: e-Vapor Product A; [analysis description as in outcome 22, analysis 1]; Test type: Equivalence — [test comment as in outcome 22, analysis 1]; p < .0001, ANOVA; Mean Difference (Net) = 0.036, 95% CI 2-sided [0.031 to 0.040]
Statistical Analysis 2: Comparison: e-Vapor Product B; [analysis description as in outcome 22, analysis 1]; Test type: Equivalence — [test comment as in outcome 22, analysis 1]; p < .0001, ANOVA; Mean Difference (Net) = 0.036, 95% CI 2-sided [0.032 to 0.041]
Statistical Analysis 3: Comparison: e-Vapor Product C; [analysis description as in outcome 22, analysis 1]; Test type: Equivalence — [test comment as in outcome 22, analysis 1]; p < .0001, ANOVA; Mean Difference (Net) = 0.041, 95% CI 2-sided [0.037 to 0.046]
Statistical Analysis 4: Comparison: e-Vapor Product D; [analysis description as in outcome 22, analysis 1]; Test type: Equivalence — [test comment as in outcome 22, analysis 1]; p < .0001, ANOVA; Mean Difference (Net) = 0.038, 95% CI 2-sided [0.033 to 0.042]

24. Secondary Outcome: Summary Statistics of Total Cartridge Weight Change by Test Product, Per Subject, During the Ad Libitum-Use Sessions
Description: Difference in recorded weight (measured in grams) by test product, per subject, collected before and after product use in ad libitum sessions
Time Frame: Samples were collected over the 12-hour ad libitum product use session on the day the subject was assigned the test product (according to the randomization scheme)
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 31
Grams | 0.534 (0.43562) | 0.406 (0.32699) | 0.469 (0.36765) | 0.418 (0.33120)
Statistical Analysis 1: Comparison: e-Vapor Product A; [analysis description as in outcome 22, analysis 1]; Test type: Equivalence — [test comment as in outcome 22, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 0.536, 95% CI 2-sided [0.407 to 0.665] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 2: Comparison: e-Vapor Product B; [analysis description as in outcome 22, analysis 1]; Test type: Equivalence — [test comment as in outcome 22, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 0.408, 95% CI 2-sided [0.280 to 0.537] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 3: Comparison: e-Vapor Product C; [analysis description as in outcome 22, analysis 1]; Test type: Equivalence — [test comment as in outcome 22, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 0.468, 95% CI 2-sided [0.339 to 0.596] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 4: Comparison: e-Vapor Product D; [analysis description as in outcome 22, analysis 1]; Test type: Equivalence — [test comment as in outcome 22, analysis 1]; p < .0001, ANCOVA; Mean Difference (Net) = 0.430, 95% CI 2-sided [0.301 to 0.559] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence

25. Secondary Outcome: Total Weight Change by Test Product and Individual Cartridge During the Ad-Libitum-Use Sessions
Description: Change in cartridge weight (measured in grams) as measured before and after a 12-hour ad-libitum use session of the product.
Time Frame: as for outcome 24
Population: Cartridges of products utilized by participants during 12-hour ad-libitum-use session
Measure: Mean (Standard Deviation); unit: Grams
Units Other Than Participants: Cartridges
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Number analyzed (Cartridges) | 42 | 39 | 39 | 35
Grams
  Cartridge 1: number analyzed (Cartridges) | 32 | 32 | 32 | 31
  Cartridge 1 | 0.428 (0.26613) | 0.310 (0.22996) | 0.398 (0.25131) | 0.369 (0.23418)
  Cartridge 2: number analyzed (Cartridges) | 8 | 6 | 6 | 4
  Cartridge 2 | 0.351 (0.25264) | 0.381 (0.24206) | 0.309 (0.26700) | 0.383 (0.21158)
  Cartridge 3: number analyzed (Cartridges) | 2 | 1 | 1 | 0
  Cartridge 3 | 0.293 (0.06010) | 0.812 (0) | 0.444 (0) |
  Overall | 0.407 (0.25716) | 0.333 (0.24023) | 0.385 (0.24910) | 0.370 (0.22882)

26. Secondary Outcome: Summary Statistics of Puff Count by Test Product During the Ad Libitum-Use Sessions
Description: Number of puffs, by test product, per subject, taken during 12-hour ad libitum product use session
Time Frame: Data was collected over the 12-hour ad libitum product use session on the day the subject was assigned the test product (according to the randomization scheme)
Measure: Mean (Standard Deviation); unit: puffs
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 31 | 32 | 31
puffs | 292.375 (204.2479) | 239.000 (164.4613) | 246.375 (170.3419) | 242.839 (194.6732)
Statistical Analysis 1: Comparison: e-Vapor Product A; Null Hypothesis: Mean Puff Count is equal to 0 Alternative Hypothesis: Mean Puff Count is not equal to 0; Test type: Equivalence — Null Hypothesis: Mean Puff Count is equal to 0 Alternative Hypothesis: Mean Puff Count is not equal to 0; p < .0001, ANCOVA; Mean Difference (Final Values) = 277.79, 95% CI 2-sided [213.62 to 341.96] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 2: Comparison: e-Vapor Product B; Null Hypothesis: Mean Puff Count is equal to 0 Alternative Hypothesis: Mean Puff Count is not equal to 0; Test type: Equivalence — Null Hypothesis: Mean Puff Count is equal to 0 Alternative Hypothesis: Mean Puff Count is not equal to 0; p < .0001, ANCOVA; Mean Difference (Final Values) = 241.32, 95% CI 2-sided [176.99 to 305.64] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 3: Comparison: e-Vapor Product C; Null Hypothesis: Mean Puff Count is equal to 0 Alternative Hypothesis: Mean Puff Count is not equal to 0; Test type: Equivalence — Null Hypothesis: Mean Puff Count is equal to 0 Alternative Hypothesis: Mean Puff Count is not equal to 0; p < .0001, ANCOVA; Mean Difference (Final Values) = 248.22, 95% CI 2-sided [184.01 to 312.43] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 4: Comparison: e-Vapor Product D; Null Hypothesis: Mean Puff Count is equal to 0 Alternative Hypothesis: Mean Puff Count is not equal to 0; Test type: Equivalence — Null Hypothesis: Mean Puff Count is equal to 0 Alternative Hypothesis: Mean Puff Count is not equal to 0; p < .0001, ANCOVA; Mean Difference (Final Values) = 257.92, 95% CI 2-sided [193.58 to 322.26] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence

27. Secondary Outcome: Average Puff Duration by Test Product During the Ad Libitum-Use Sessions
Description: Seconds per puff taken, by test product, per subject, during 12-hour ad libitum product use session
Time Frame: as for outcome 26
Measure: Mean (Standard Deviation); unit: seconds per puff
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 31 | 30 | 31 | 30
seconds per puff | 2.471 (1.01786) | 2.373 (1.10711) | 2.249 (0.89143) | 2.209 (0.75672)
Statistical Analysis 1: Comparison: e-Vapor Product A; Null Hypothesis: Mean Average Puff Duration is equal to 0 Alternative Hypothesis: Mean Average Puff Duration is not equal to 0; Test type: Equivalence — Null Hypothesis: Mean Average Puff Duration is equal to 0 Alternative Hypothesis: Mean Average Puff Duration is not equal to 0; p < .0001, ANCOVA; Mean Difference (Final Values) = 2.223, 95% CI 2-sided [1.915 to 2.580] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 2: Comparison: e-Vapor Product B; [analysis description as in outcome 27, analysis 1]; Test type: Equivalence — [test comment as in outcome 27, analysis 1]; p < .0001, ANCOVA; Mean Difference (Final Values) = 2.203, 95% CI 2-sided [1.897 to 2.557] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 3: Comparison: e-Vapor Product C; [analysis description as in outcome 27, analysis 1]; Test type: Equivalence — [test comment as in outcome 27, analysis 1]; p < .0001, ANCOVA; Mean Difference (Final Values) = 2.101, 95% CI 2-sided [1.810 to 2.439] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 4: Comparison: e-Vapor Product D; [analysis description as in outcome 27, analysis 1]; Test type: Equivalence — Null Hypothesis: Mean Total Puff Duration is equal to 0 Alternative Hypothesis: Mean Total Puff Duration is not equal to 0; p < .0001, ANCOVA; Mean Difference (Final Values) = 2.052, 95% CI 2-sided [1.767 to 2.382] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence

28. Secondary Outcome: Total Puff Duration by Test Product During the Ad Libitum-Use Sessions
Description: Total seconds puffing by test product, per subject, taken during 12-hour ad libitum product use session
Time Frame: as for outcome 26
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 31 | 30 | 31 | 30
Seconds | 726.028 (551.0662) | 589.204 (435.7242) | 575.807 (442.4253) | 517.733 (386.5348)
Statistical Analysis 1: Comparison: e-Vapor Product A; Null Hypothesis: Mean Total Puff Duration is equal to 0 Alternative Hypothesis: Mean Total Puff Duration is not equal to 0; Test type: Equivalence — [test comment as in outcome 27, analysis 4]; p < .0001, ANCOVA; Mean Difference (Final Values) = 709.86, 95% CI 2-sided [549.19 to 870.54] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 2: Comparison: e-Vapor Product B; [analysis description as in outcome 28, analysis 1]; Test type: Equivalence — [test comment as in outcome 27, analysis 4]; p < .0001, ANCOVA; Mean Difference (Final Values) = 568.35, 95% CI 2-sided [407.18 to 729.51] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 3: Comparison: e-Vapor Product C; [analysis description as in outcome 28, analysis 1]; Test type: Equivalence — [test comment as in outcome 27, analysis 4]; p < .0001, ANCOVA; Mean Difference (Final Values) = 562.00, 95% CI 2-sided [401.34 to 722.67] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence
Statistical Analysis 4: Comparison: e-Vapor Product D; [analysis description as in outcome 28, analysis 1]; Test type: Equivalence — [test comment as in outcome 27, analysis 4]; p < .0001, ANCOVA; Mean Difference (Final Values) = 517.23, 95% CI 2-sided [356.11 to 678.34] — LSM calculated from mixed models. Each model includes fixed effect terms for product, period and sequence

29. Secondary Outcome: Total Cartridges Used by Test Product During the Ad Libitum-Use Sessions
Description: Total cartridges used by test product, per subject, taken during 12-hour ad libitum product use session
Time Frame: as for outcome 26
Measure: Mean (Standard Deviation); unit: Cartridges
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 31
Cartridges | 1.313 (0.59229) | 1.219 (0.49084) | 1.219 (0.49084) | 1.129 (0.34078)

30. Secondary Outcome: Summary of Binary VAS-Derived Categorical "Use Product Again Questionnaire" Scores by Test Product
Description: Visual Analog Scale (VAS) measuring self-reported response to "Use the product again" questionnaire was collected after each product use session. The questionnaire consists of a single question ("If given the opportunity, I would want to use this product again"). Participants indicated their willingness to use the product again by pointing to a line measuring 100mm, with scores measured from left to right and ranging between 0 to 100 mm. Scores closer to the right, and thus higher on the scale, indicated a greater willingness to utilize the product again. Raw scores were converted to a binary score as follows: VAS scores < 50 mm ≈ unwillingness to use the product again, and VAS scores ≥ 50 mm ≈ willingness to use product again.
Time Frame: Data was collected at the end of the 12-hour ad libitum product use session on the day the subject was assigned the test product (according to the randomization scheme)
Measure: Count of Participants; unit: Participants
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants
  Want to Use | 29 | 29 | 27 | 28
  Do not Want to Use | 3 | 3 | 5 | 4

31. Secondary Outcome: Summary of Ordinal VAS-Derived Categorical "Use Product Again Questionnaire" Scores by Test Product
Description: Visual Analog Scale (VAS) measuring self-reported response to willingness to use study product again. Questionnaire was collected after each product use session. Questionnaire consists of a single question ("If given the opportunity, I would want to use this product again") with VAS response range from "Definitely Would Not" to "Don't Care" to "Definitely Would". Participants indicated their willingness to use the product again by pointing to a line measuring 100mm, with scores measured from left to right and ranging between 0 to 100 mm. Scores closer to the right, and thus higher on the scale, indicated a greater willingness to utilize the product again. The raw scores were then converted to a binary, "unwilling" vs. "willing" to use response. Additionally, a 3-level ordinal response was computed using "unwilling" (VAS < 50 mm), "don't care" (VAS = 50 mm), and "willing" (VAS > 50 mm).
Time Frame: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Participants
  Want to Use | 29 | 29 | 26 | 28
  Don't Care | 0 | 0 | 1 | 0
  Do Not Want to Use | 3 | 3 | 5 | 4

32. Secondary Outcome: Puff Count by Test Product and Individual Cartridge During the Ad-Libitum-Use Sessions
Description: Puff Count by Test Product (Pooled Over Cartridges) during 12-hour ad-libitum-use session of the product.
Time Frame: Over the 12-hour ad libitum product use session on the day the subject was assigned the test product (according to the randomization scheme)
Population: Cartridges of products utilized by participants during 12-hour ad-libitum-use session
Measure: Mean (Standard Deviation); unit: Puffs
Units Other Than Participants: Cartridges
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Number analyzed (Cartridges) | 42 | 37 | 39 | 35
Puffs
  Cartridge 1: number analyzed (Cartridges) | 32 | 31 | 32 | 31
  Cartridge 1 | 247.156 (146.7016) | 197.065 (147.5464) | 217.969 (143.7912) | 220.032 (141.3675)
  Cartridge 2: number analyzed (Cartridges) | 8 | 5 | 6 | 4
  Cartridge 2 | 164.250 (121.5680) | 195.600 (98.79929) | 117.333 (130.9712) | 176.750 (193.3190)
  Cartridge 3: number analyzed (Cartridges) | 2 | 1 | 1 | 0
  Cartridge 3 | 66.500 (27.57716) | 322.000 (0) | 205.000 (0) |
  Overall | 222.762 (145.3878) | 200.243 (140.1773) | 202.154 (143.0770) | 215.086 (145.3491)

33. Secondary Outcome: Average Puff Duration by Test Product and Individual Cartridge During the Ad-Libitum-Use Sessions
Description: Average puff duration (measured in seconds) by Test Product (Pooled Over Cartridges) during 12-hour ad-libitum-use session of the product.
Time Frame: as for outcome 32
Population: Cartridges of products utilized by participants during 12-hour ad-libitum-use session
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Cartridges
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Number analyzed (Cartridges) | 41 | 36 | 37 | 34
Seconds
  Cartridge 1: number analyzed (Cartridges) | 31 | 30 | 31 | 30
  Cartridge 1 | 2.487 (1.05031) | 2.369 (1.10274) | 2.275 (0.92685) | 2.194 (0.73162)
  Cartridge 2: number analyzed (Cartridges) | 8 | 5 | 5 | 4
  Cartridge 2 | 2.674 (1.13172) | 3.111 (1.52758) | 3.004 (0.89069) | 2.685 (1.32845)
  Cartridge 3: number analyzed (Cartridges) | 2 | 1 | 1 | 0
  Cartridge 3 | 4.761 (0.06038) | 3.598 (0) | 3.330 (0) |
  Overall | 2.634 (1.13792) | 2.506 (1.17333) | 2.402 (0.94449) | 2.252 (0.81028)

34. Secondary Outcome: Total Puff Duration by Test Product and Individual Cartridge During the Ad-Libitum-Use Sessions
Description: Total Puff Duration (measured in seconds) by Test Product (pooled over cartridges) during 12-hour ad-libitum-use session of the product.
Time Frame: as for outcome 32
Population: Cartridges of products utilized by participants during 12-hour ad-libitum-use session
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Cartridges
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 32 | 32 | 32 | 32
Number analyzed (Cartridges) | 41 | 36 | 37 | 34
Seconds
  Cartridge 1: number analyzed (Cartridges) | 31 | 30 | 31 | 30
  Cartridge 1 | 597.673 (366.5793) | 455.996 (299.0212) | 486.874 (274.7173) | 463.815 (273.8106)
  Cartridge 2: number analyzed (Cartridges) | 8 | 5 | 5 | 4
  Cartridge 2 | 418.433 (293.8095) | 567.524 (247.0947) | 414.832 (411.0123) | 404.380 (352.2326)
  Cartridge 3: number analyzed (Cartridges) | 2 | 1 | 1 | 0
  Cartridge 3 | 315.777 (127.2806) | 1158.612 (0) | 682.752 (0) |
  Overall | 548.948 (352.5085) | 491.003 (309.3294) | 482.433 (288.8387) | 456.823 (278.4626)

35. Secondary Outcome: Total Weight Change by Test Product, Per Completed Cartridge, During the Ad-Libitum-Use Sessions
Description: as for outcome 25
Time Frame: as for outcome 32
Population: Cartridges of products utilized by participants during 12-hour ad-libitum-use session
Measure: Mean (Standard Deviation); unit: Grams
Units Other Than Participants: Cartridges
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 8 | 6 | 6 | 5
Number analyzed (Cartridges) | 10 | 7 | 7 | 5
Grams | 0.623 (0.24705) | 0.315 (0.18197) | 0.664 (0.19375) | 0.656 (0.15309)

36. Secondary Outcome: Average Puff Duration by Test Product, Per Completed Cartridge, During the Ad-Libitum-Use Sessions
Description: Average puff duration (measured in seconds) by Test Product, per completed cartridge, during a 12-hour ad-libitum use session of the product.
Time Frame: as for outcome 32
Population: Cartridges of products utilized by participants during 12-hour ad-libitum-use session
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Cartridges
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 8 | 6 | 6 | 5
Number analyzed (Cartridges) | 10 | 7 | 7 | 5
Seconds | 3.033 (1.30359) | 3.004 (1.27635) | 3.019 (0.93719) | 2.491 (0.60612)

37. Secondary Outcome: Puff Count by Test Product, Per Completed Cartridge, During the Ad-Libitum-Use Sessions
Description: Puff count by Test Product, per completed cartridge, during a 12-hour ad-libitum use session of the product.
Time Frame: as for outcome 32
Population: Cartridges of products utilized by participants during 12-hour ad-libitum-use session
Measure: Mean (Standard Deviation); unit: Puffs
Units Other Than Participants: Cartridges
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 8 | 6 | 6 | 5
Number analyzed (Cartridges) | 10 | 7 | 7 | 5
Puffs | 298.300 (155.1444) | 159.714 (108.9567) | 280.000 (137.6311) | 311.400 (171.0111)

38. Secondary Outcome: Total Puff Duration by Test Product, Per Completed Cartridge, During the Ad-Libitum-Use Sessions
Description: Total Puff Duration (measured in seconds) by Test Product, per completed cartridge, during a 12-hour ad-libitum use session of the product.
Time Frame: as for outcome 32
Population: Cartridges of products utilized by participants during 12-hour ad-libitum-use session
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Cartridges
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D
Number analyzed (Participants) | 8 | 6 | 6 | 5
Number analyzed (Cartridges) | 10 | 7 | 7 | 5
Seconds | 814.728 (350.9879) | 432.943 (240.6142) | 766.922 (307.3669) | 729.328 (317.4452)

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) data collected for entire study duration: approximately 34 days from Visit 1 (screening) through End of Study for each individual subject.
Description: Review of adverse events conducted by study staff at each study visit and documented in both source documentation and electronic Case Report Form.
Groups:
- Day -1 Product Trial Non-randomized Subjects: Subjects who were not randomized after participating in the Day -1 Product Trial using all study products including:
  Product XL25F = Test e-vapor product (EVP) (formerly marketed by Nu Mark LLC as MarkTen® XL Fusion [2.5% nicotine by weight {NBW}]) e-Vapor Product A: e-Vapor product Product XL40CB = Test EVP (formerly marketed by Nu Mark LLC as MarkTen® XL Bold Classic [4.0% NBW]) e-Vapor Product B: e-Vapor product Product XL35WM = Test EVP (formerly marketed by Nu Mark LLC as MarkTen® XL Winter Mint [3.5% NBW] e-Vapor Product C: e-Vapor product Product XL40MB = Test EVP (formerly marketed by Nu Mark LLC as MarkTen® XL Bold Menthol [4.0% NBW]) e-Vapor Product D: e-Vapor product
Arm/Group | e-Vapor Product A | e-Vapor Product B | e-Vapor Product C | e-Vapor Product D | Day -1 Product Trial Non-randomized Subjects
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32 | 0/3
Other Adverse Events (participants affected / at risk) | 3/32 | 1/32 | 3/32 | 4/32 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | e-Vapor Product A (N=32) | e-Vapor Product B (N=32) | e-Vapor Product C (N=32) | e-Vapor Product D (N=32) | Day -1 Product Trial Non-randomized Subjects (N=3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Coughing

LIMITATIONS AND CAVEATS:
In this study, a cut off of greater than 50% of the samples too low to be detected was used to determine which analytes would be analyzed with a mixed model. Exhaled acetaldehyde and acrolein amounts were not detectable in 100% of subjects; therefore the differences in concentrations between sham and product trials for these analytes were not analyzed as intended in the statistical analysis plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04881942/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT04881942/SAP_001.pdf